CLINICAL TRIAL: NCT01144117
Title: Double Blind, Placebo-controlled Study to Assess the Effects of Erythropoietin on Clinical Disability and Brain Pathology as Shown by Magnetic Resonance Imaging in Patients With Progressive Multiple Sclerosis
Brief Title: The Effects of Erythropoietin on Clinical Disability and Brain Pathology in Patients With Progressive Multiple Sclerosis
Acronym: EPO-ProgMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Research Centre for Magnetic Resonance (Other)
Responsible Party: Professor Per Soelberg Sorensen, Rigshospitalet., The Danish MS Research Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT number: 2009-011516-37
Record Dates: First submitted 2010-06-07; First posted 2010-06-15 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2010-05

CONDITIONS: Multiple Sclerosis (Primary or Secondary Progressive Phase).
Keywords: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Erythropoietin; Eosinophil Peroxidase; epoetin beta

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erythropoietin (Experimental): Erythropoietin treated patients contra placebo.
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — Erythropoietin 48000 IU given I.V. in 17 courses
  Other Names: Epo, NeoRecormon

SUMMARY:
In a double-blind, placebo-controlled, parallel group trial, recombinant human erythropoietin (rhEPO) (48000 IU) treatment or placebo will be administered weekly i.v. for 24 weeks: weekly for 12 weeks and bi-weekly for 12 weeks. Methylprednisolone (MP) 1 g i.v. will be administered before the first and second EPO/placebo administration. The 24-week treatment period will be followed by a 24-week observation period.

DETAILED DESCRIPTION:
Patients with primary progressive MS or secondary progressive MS without relapses during the last 1 year will be suitable for the trial. In all 56 patients will be enrolled into the study.

The primary outcome measure is the change from baseline to 24 weeks in a composite of maximum gait distance, 9-hole peg test, TRAIL making B comparing the placebo-treatment group with the EPO-treatment group.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 60 years
* primary progressive MS or secondary progressive MS without relapses during the last one year
* duration of the disease of at least 2 years Clinical disability progression should have been observed in the 2 years prior to screening as per clinical judgment of the investigator. In addition, progression must be documented by an increase in the EDSS score of at least 0.5 points at any time during the 2 years prior to Screening; or progression of 1 point in the pyramidal, cerebellar, brain stem , visual or sensory functional system during the last 2 years. Should documented EDSS scores not be available, a written summary of the clinical evidence of disability progression in the previous 2 years must be submitted (for example walking distance or hand function).
* EDSS (Expanded Disability Status Scale) 4.0-6.5
* MRI fulfilling the Barkhof criteria for MS
* written informed consent

Exclusion Criteria:

* pregnancy or period of breastfeeding or missing adequate contraceptive protection
* treatment with steroids in the last 30 days
* treatment with interferons, glatiramer acetate or IVIG in the last1 month prior to enrolment
* treatment with azathioprin, mitoxantrone or any other immuno-suppressive in the 6 months prior to enrolment
* cardiac insufficiency (NYHA III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, instable or advanced ischemic heart disease (CCS III or IV), malignant hypertension (systolic > 180, diastolic > 110)
* history of any haematological disorder
* history of renal insufficiency
* any medical psychiatric or other circumstances which impede or restrict the subjects participation in the study in the manner intended
* contraindication for contrast enhanced MRI (e.g. pace maker, aortic clip or any metal implant)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the change from baseline to 24 weeks in a composite of maximum gait distance, 9-hole peg test, TRAIL making B comparing the placebo-treatment group with the EPO-treatment group. | 48 weeks

SECONDARY OUTCOMES:
Comparisons between the placebo-and the EPO-group regarding:difference in maximum gait distance between baseline and week 24. | 48 weeks
Comparisons between the placebo-and the EPO-group regarding:difference in 9-hole peg test | 48 weeks
Comparisons between the placebo-and the EPO-group regarding:difference in TRAIL making B | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Schreiber, MD., Ph.d., Principal Investigator — Rigshospitalet, Denmark; Per S Soerensen, MD., Prof, Study Director — Rigshospitalet, Denmark
Locations (1):
- Karen Schreiber, Copenhagen, Oesterbro, Denmark